CLINICAL TRIAL: NCT00442182
Title: The Effects and Side Effects of ITS2357 in Autoinflammatory Syndromes
Brief Title: The Efficacy and Safety of ITF2357 in AIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/112
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Autoinflammatory Syndromes; HIDS; TRAPS; Schnitzler's Syndrome
Keywords: autoinflammatory syndromes
MeSH Terms: conditions — Schnitzler Syndrome | interventions — givinostat hydrochloride

INTERVENTIONS:
Drug: ITF2357

SUMMARY:
Autoinflammatory syndromes (AIS) are a group of disorders characterized by recurrent episodes of inflammation.Although for the hereditary autoinflammatory diseases the genetic mutations are known it remains largely unclear how these mutations lead to recurrent inflammatory attacks. Treatment of the inflammatory symptoms remains a challenge. With beneficial responses reported during treatment with simvastatin, etanercept or anakinra in some but not all patients. ITF2357 is an orally active histon deacetylase inhibitor with a potent anti-inflammatory effect due to inhibition of pro-inflammatory cytokines (IL-1β, TNFα, IFNg, IL-6). We expect that ITF2357 is able to modify the clinical symptoms of AIS patients and induce clinical complete remission or a reduction in attack duration.

DETAILED DESCRIPTION:
Rationale: Autoinflammatory syndromes (AIS) are a group of disorders characterized by recurrent episodes of inflammation. This occurs in the absence of autoantibodies and antigen specific T cells. To date 6 genetically distinct hereditary autoinflammatory syndromes are known and more recently other sporadic syndromes, such as the Schnitzler's syndrome (urticaria, periodic fever and paraproteinemia) and Periodic Fever Aphtous stomatitis, Pharyngitis and Adenitis (PFAPA) are being recognized as AIS. Amyloidosis is a serious complication of chronic or recurrent inflammation seen in some of these syndromes. Although for the hereditary autoinflammatory diseases the genetic mutations are known it remains largely unclear how these mutations lead to recurrent inflammatory attacks. Symptomatic episodes are associated with increased serum concentrations of both pro-inflammatory mediators (TNFα, IL-6, IL1β and IFN-g) as well as of the anti-inflammatory compounds (IL-1ra, sTNFR p55 and sTNFR p75). In vitro and ex vivo experiments suggest a central role in the pathogenesis for IL-1β. The observation that rIL-1ra (anakinra) is highly effective in refractory TRAPS, CAPS, HIDS, refractory FMF and SS support this idea. Despite its effectiveness daily painful subcutaneous injections and injection site reactions remain a problem. ITF2357 is an orally active histon deacetylase inhibitor with a potent anti-inflammatory effect due to inhibition of pro-inflammatory cytokines (IL-1β, TNFα, IFNg, IL-6). We expect that ITF2357 is able to modify the clinical symptoms of AIS patients and induce clinical complete remission or a reduction in attack duration.

Objective: The primary objective is to asses whether ITF2357 is able to induce clinical complete remission in patients with continuous symptoms or reduce attack duration with > 33% in periodically symptomatic patients. Secondary objectives are the emergence of adverse events and toxicity as well as the influence of ITF2357 on cytokine production and laboratory parameters for infection and metabolism.

Study design: Open Label Pilot Study Study population: AIS patients 18 years or older with severe disease

Intervention: Patients with continuous symptoms will receive 2-3 times a day 50mg (capsule) ITF2357 for a total period of 90 days. Patients with periodic symptoms will take ITF2357 (2-3 times a day 50mg) on 7-14 consecutive days during 6-12 attacks.

Main study parameters: A clinical complete remission will be regarded as a clinical score (CS) < 10 scored on the symptom score list in the absence of a temperature > 38.0°C and normalisation of CRP and WBC levels. The end of an attack will be defined as a CS < 20 in the absence of a temperature > 38.0°C.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients will be admitted once at the beginning of the study for 3 days in this period there will be performed a daily venipuncture, a history and physical examination twice and an ECG once. They will visit the outpatient clinic four times for physical examination, history, venipuncture and an ECG. Patients are asked to complete a symptom score list on which they can note down the date, number of ITF2357 capsules taken and if present co-medication, symptoms, temperature and adverse events. Patients are asked to collect a portion of morning urine once a week. ITF2357 showed the following adverse reactions asymptomatic trombocytopenia and perhaps increased incidence of mild infections mainly of the upper respiratory tract. There were gastrointestinal complaints in the sense of nausea, vomiting, abdominal pain and diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Autoinflammatory syndrome (hereditary or acquired)
* Age ³18 years
* Severe active disease (≥1 attack every eight weeks or continuous symptoms).

An attack will be defined as:

* Temperature of ≥38 ºC not otherwise explained.
* At least two other accompanying symptoms (e.g. joint pain, lymphadenopathy, skin lesions, abdominal symptoms)
* written informed consent obtained

Exclusion Criteria:

* Age < 18 years
* Pregnancy and lactation
* Increased risk for infection or current infection
* Renal failure (GFR<30ml/1.73m2/min)
* Pre-existing malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-09

PRIMARY OUTCOMES:
clinical complete remission
number of days of illness

SECONDARY OUTCOMES:
side effects

CONTACTS AND LOCATIONS:
Overall Officials: Jos WM van der Meer, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre Nijmegen, Nijmegen, Netherlands